CLINICAL TRIAL: NCT00592813
Title: Efficacy of a Post-Rehabilitation Exercise Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Alan Jette, Director, Health and Disability Research Institute, Boston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NINR 1R01NR010815-01A2; 1R01NR010815-01A2 (NIH)
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Hip Fracture; Disability
Keywords: rehabilitation; function
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Enhanced Strong for Life
- cardiovascular education (attention control) (Placebo Comparator)
  Interventions: Behavioral: cardiovascular nutrition education

INTERVENTIONS:
Behavioral: Enhanced Strong for Life — The program contains 5 minutes of warm-up, 25 minutes of strengthening, and 5 minutes of cool-down exercises. The SFL program is contained on a 35 minute videotape. Subjects are instructed to increase resistance when they can perform 10 repetitions of a movement pattern without significant fatigue or loss of proper execution. Subjects are instructed to move within a comfortable range of motion.
  Participants will be taught the SFL program during two home visits conducted by a physical therapist. On the first visit, the exercise techniques will be taught, modified as needed based on individual needs and practiced as necessary until proper technique is attained. Each participant will be given written guidelines for how to progress resistance of the program, how to modify the exercises and how to complete bimonthly exercise calendars.
  Arms: 1
Behavioral: cardiovascular nutrition education — administered as an attention control intervention using home visits, phone calls and mail-outs of information
  Arms: cardiovascular education (attention control)

SUMMARY:
Background:

Many people who have suffered a hip fracture are discharged from rehabilitation services with significant residual functional limitations and disability. We believe that a home-based exercise program that incorporates cognitive-behavioral techniques to increase exercise adherence and promote the return to daily activities could extend the benefits of formal rehabilitation for patients who have suffered a hip fracture.

Specific Aims:

We will conduct a 5-year multi-site randomized controlled trial in patients who have suffered a recent hip fracture and have completed all rehabilitation services. The specific aim that this project will address is whether:

Participation in the Strong for Life (SFL) program will improve function and disability outcomes in participants 6-months after they are discharged from rehabilitation services.

This study will also investigate the following secondary hypotheses:

1. Changes in function and disability at 6-month follow-up will be correlated with changes in all three proposed intermediary variables: muscle strength, balance, and self-efficacy.
2. The SFL program will significantly improve health-related quality of life among participants at 6-month follow-up.
3. At 9-month follow-up the SFL program will continue to have a significant impact on participants' function and disability compared to the control group.

Target population:

The target population will be people aged 60 years or more who have suffered a recent traumatic hip fracture, have one or more residual functional limitations and have completed all inpatient, outpatient or homecare rehabilitation services.

Intervention:

We will use an enhanced version of the Strong for Life program. This home-based exercise program will include both resistance exercises using Thera-bands that will be shown on a video/DVD and weight-bearing exercises that are progressed using a step and/or a weighted vest. A cognitive-behavioral program that is customized for people recovering from hip fracture is being developed that will focus on promoting exercise adherence, decreasing fear of falling and increasing the return to daily activities in the patient's home and community.

Design:

A randomized controlled clinical trial will be implemented to measure the efficacy of the Strong for Life program. An attention-control intervention will be provided to all participants assigned to the control group. The outcome evaluation points are:

* T0: baseline, at the point of discharge from formal rehabilitation;
* T2: 6-month outcome assessment
* T3: 9-month follow-up

Outcomes:

The primary outcomes will be function measured by both self-report (AM PAC) and physical performance measures (SPPB). Secondary outcomes include disability, self-efficacy, balance, strength, cognition, and reaction time. Adherence to the exercise program and adverse events will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Have a primary diagnosis of hip fracture;
* Aged 60 years and above;
* Have functional limitation (i.e., as determined by limitation in at least one of 9 functional tasks listed in the SF-36 physical function scale, excluding vigorous activities);
* Have recently been discharged from rehabilitation services;
* Be able to understand and communicate in English;
* Be able to safely and independently stand with or without the aid of a mobility device, without needing any assistance or supervision from another person;
* Have received written clearance from their primary care physician documenting no contra-indications for participating in the study;
* Be able to provide written informed consent.

Exclusion Criteria:

* Have serious cognitive deficits (i.e., a Mini-Mental State Examination score of less than 20)85;
* Have severe depression (i.e., a score of 20 or greater on the Geriatric Depression Scale)86;
* Have a terminal illness with survival expected to be less than 1 year;
* Have significant pulmonary or cardiovascular contraindications or pre-existing conditions that preclude participating in an exercise program;
* Legally blind;
* Currently receiving rehabilitation therapy;
* Live outside of the study's catchment area in the Boston metropolitan area and eastern Massachusetts.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2008-04; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The specific aim that this project will address is whether: Participation in the SFL program will improve function and disability outcomes in participants 6-months after they are discharged from rehabilitation services. | baseline, 6-month and 9-month follow up
  performance based function is assessed using the Short Physical Performance Battery (SPPB) and self-reported function is assessed using the AM-PAC

SECONDARY OUTCOMES:
Changes in function and disability at 6-month follow-up will be correlated with changes in all three proposed intermediary variables: muscle strength, balance, and self-efficacy. | baseline, 6-month and 9-month follow up
At 9-month follow-up the SFL program will continue to have a significant impact on participants' function and disability compared to the control group. | baseline, 6-month and 9-month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Alan M Jette, PhD, Principal Investigator — Health & Disability Research Institute; Nancy Latham, PhD, Principal Investigator — Health & Disability Research Institute
Locations (1):
- Spaulding Rehabilitation Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Latham NK, Harris BA, Bean JF, Heeren T, Goodyear C, Zawacki S, Heislein DM, Mustafa J, Pardasaney P, Giorgetti M, Holt N, Goehring L, Jette AM. Effect of a home-based exercise program on functional recovery following rehabilitation after hip fracture: a randomized clinical trial. JAMA. 2014 Feb 19;311(7):700-8. doi: 10.1001/jama.2014.469. PMID 24549550